CLINICAL TRIAL: NCT05483933
Title: An Open-Label, Phase 1b Study of SL-172154 (SIRPα-Fc-CD40L) Administered With Either Pegylated Liposomal Doxorubicin or Mirvetuximab Soravtansine in Subjects With Platinum-Resistant Ovarian Cancers
Brief Title: Phase 1b Study of SL-172154 Administered With Combination Agent(s) in Subjects With Ovarian Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shattuck Labs, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SL03-OHD-105
Record Dates: First submitted 2022-07-26; First posted 2022-08-02 (Actual); Results first posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Platinum-resistant Ovarian Cancer; Fallopian Tube Cancer; Epithelial Ovarian Cancer; Ovarian Cancer; Platinum-Resistant Fallopian Tube Carcinoma; Platinum-Resistant Primary Peritoneal Carcinoma; Primary Peritoneal Carcinoma
Keywords: Platinum-resistant; Ovarian; Peritoneal; High grade serous EOC; primary peritoneal cancer; Fallopian; Combination; Mirvetuximab Soravtansine; SL-172154; SIRPα-Fc-CD40L; Pegylated Liposomal Doxorubicin
MeSH Terms: conditions — Fallopian Tube Neoplasms; Carcinoma, Ovarian Epithelial; Ovarian Neoplasms | interventions — liposomal doxorubicin; 1-dodecylpyridoxal; mirvetuximab soravtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pegylated Liposomal Doxorubicin + SL-172154 (SIRPα-Fc-CD40L) (Experimental): Pegylated Liposomal Doxorubicin (PLD) will be administered via intravenous administration + SL-172154 (SIRPα-Fc-CD40L) will be administered via intravenous administration.
  Interventions: Drug: Pegylated Liposomal Doxorubicin + SL-172154
- Mirvetuximab + SL-172154 (SIRPα-Fc-CD40L) (Experimental): Mirvetuximab (MIRV) will be administered via intravenous administration + SL-172154 (SIRPα-Fc-CD40L) will be administered via intravenous administration
  Interventions: Drug: Mirvetuximab + SL-172154

INTERVENTIONS:
Drug: Pegylated Liposomal Doxorubicin + SL-172154 — The investigational product, SL-172154, is a novel fusion protein consisting of human SIRPα and CD40L (SIRPα -Fc-CD40L) linked via a human Fc.
  Other Names: Doxil; PLD; Caelyx
  Arms: Pegylated Liposomal Doxorubicin + SL-172154 (SIRPα-Fc-CD40L)
Drug: Mirvetuximab + SL-172154 — The investigational product, SL-172154, is a novel fusion protein consisting of human SIRPα and CD40L (SIRPα -Fc-CD40L) linked via a human Fc.
  Other Names: IMGN853; MIRV
  Arms: Mirvetuximab + SL-172154 (SIRPα-Fc-CD40L)

SUMMARY:
SL03-OHD-105 is an open-label, multicenter, phase 1b trial designed to evaluate SL-172154 administered in combination with pegylated liposomal doxorubicin (PLD) or mirvetuximab soravtansine (MIRV) in patients with platinum resistant ovarian cancer. Approximately 102 patients will be enrolled in this study.

DETAILED DESCRIPTION:
Study SL03-OHD-105 is an open-label, multicenter, phase 1b trial designed to evaluate the safety, pharmacokinetics, pharmacodynamic effects, and preliminary anti-tumor activity of SL-172154 administered in combination with either PLD or MIRV in subjects with platinum-resistant ovarian, primary peritoneal, or fallopian tube cancers. Patients will be appropriate for combination therapy for their next line of therapy. For the SL-172154 + MIRV cohort, patients' tumors must be positive (defined as PS2+ ≥ 25%) for folate receptor alpha (FRα) as defined by the Ventana FOLR1 (Folate Receptor 1/Folate Receptor Alpha) Assay.

The first portion of the study will evaluate the safety of increasing dose levels of SL-172154 in combination with either PLD or MIRV and establish a combination dose for both regimens to be further evaluated in two dose expansion cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has voluntarily agreed to participate by giving written informed consent in accordance with ICH/GCP guidelines and applicable local regulations.
2. Age ≥18 years
3. [PLD Cohort] Subject has a histologically confirmed diagnosis of high grade epithelial ovarian cancer, including primary peritoneal cancer or fallopian tube cancer. Non-epithelial tumors and ovarian tumors with low malignant potential are excluded.
4. [PLD Cohort] Subject must have platinum-resistant disease, defined as radiologic disease progression within 180 days (6 months) following the last administered dose of platinum therapy. Subjects who are primary platinum-refractory, defined by progressing during or within 1 month of upfront platinum therapy, are excluded.
5. [PLD Cohort] Subjects may have received any number of prior lines of therapy for epithelial ovarian cancer; however, they may not have received more than 1 prior line of systemic anticancer therapy for platinum-resistant disease.
6. [MIRV Cohort] Subject has a histologically confirmed diagnosis of high grade serous epithelial ovarian cancer, including primary peritoneal cancer or fallopian tube cancer. Non-epithelial tumors and ovarian tumors with low malignant potential are excluded.
7. [MIRV Cohort] Subject must have platinum-resistant disease as defined by:

   * Subjects who have only had 1 line of platinum-based therapy must have received at least 4 cycles of platinum, must have had a response (complete response/remission [CR] or partial response/remission [PR]) and then progressed between >3 months and ≤6 months after the date of the last dose of platinum.
   * Subjects who have received 2 or 3 lines of platinum therapy must have progressed on or within 6 months after the date of the last dose of platinum.
   * Subjects who are platinum refractory during front-line treatment are excluded [primary platinum-refractory disease, defined as disease that did not respond to (CR or PR) or has progressed within 3 months of the last dose of first-line platinum-containing chemotherapy]
8. [MIRV Cohort] Subjects must have received at least 1 but no more than 3 prior systemic lines of anticancer therapy.
9. [MIRV Cohort] Willing to provide an archival tumor tissue block or slides or undergo procedure to obtain new biopsy using a low-risk, medically routine procedure for IHC confirmation of FRα positivity.
10. [MIRV Cohort] Subject's tumor must be positive for FRα expression (defined as PS2+ ≥ 25% by the Ventana FOLR1 Assay).
11. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1.
12. Measurable disease by RECIST v1.1 using radiologic assessment.
13. Adequate organ and hematologic function
14. Subjects must have stabilized or recovered (Grade 1 or baseline) from all prior anti-cancer therapy-related toxicities.
15. [MIRV Cohort, Dose Expansion only] Willing to consent to 1 mandatory pre-treatment and 1 on-treatment tumor biopsy, unless there is excessive risk from the procedure as determined by the investigator

Exclusion Criteria:

1. Prior treatment with a signal-regulatory protein alpha (SIRPα) targeting agent, anti-CD47 agent or CD40 agonist.
2. [PLD Cohort] Prior treatment with doxorubicin or PLD
3. [MIRV Cohort] Prior treatment with MIRV or another FRα-targeting agent
4. Any anti-cancer therapy within the time intervals specified per protocol.
5. Concurrent chemotherapy, immunotherapy, biologic or hormonal therapy for cancer treatment is prohibited.
6. Receipt of live attenuated vaccine (including live attenuated vaccines for COVID-19) within 28 days of the first dose of study treatment.
7. Current or prior use of systemic immunosuppressive medication within 7 days prior to first dose of study treatment.
8. [MIRV Cohort] Requires use of folate-containing supplements (e.g., folate deficiency)
9. Active or documented history of autoimmune disease that has required treatment with a disease modifying agent or immunosuppressive therapy in the past two years, history of multiple sclerosis (MS) or other demyelinating disease and/or Lambert-Eaton syndrome (paraneoplastic syndrome). Exceptions include controlled Type I diabetes, vitiligo, alopecia areata or hypo/hyperthyroidism.
10. Ongoing or active infection (e.g., no systemic antimicrobial therapy for treatment of infection within 5 days of D1 of study treatment).
11. Known severe hypersensitivity to the active drug substance or to any of the excipients for the agents to be administered or known hypersensitivity to Chinese hamster ovary cell products.
12. Severe gastrointestinal conditions.
13. Clinically significant or uncontrolled cardiovascular disease
14. [MIRV Cohort] History of cirrhotic liver disease (Child-Pugh Class B or C)
15. [MIRV Cohort] Active or chronic corneal disorders, history of corneal transplantation, or active ocular conditions requiring ongoing treatment/monitoring, such as uncontrolled glaucoma, wet age-related macular degeneration requiring intravitreal injections, active diabetic retinopathy with macular edema, macular degeneration, presence of papilledema, and/or monocular vision.
16. Previous clinical diagnosis of noninfectious interstitial lung disease (ILD), including noninfectious pneumonia.
17. Untreated central nervous system or leptomeningeal metastases.
18. Another malignancy that requires active therapy and that, in the opinion of the investigator and Sponsor, would interfere with monitoring of radiologic assessments of response to the study treatment.
19. Has undergone allogeneic stem cell transplantation or organ transplantation.
20. Known history or positive test for human immunodeficiency virus (HIV), or positive test for hepatitis B (positive for hepatitis B surface antigen [HBsAg]) or hepatitis C virus ([HCV]

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2022-08-18 (Actual); Primary Completion 2025-02-07 (Actual); Study Completion 2025-02-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (5):
  - University of Arkansas for Medical sciences, Little Rock, Arkansas
  - City of Hope, Duarte, California
  - Robert H.Lurie ComprehensiveCancer Center, Northwestern University, Chicago, Illinois
  - START Midwest, Grand Rapids, Michigan
  - Stephenson Cancer Center, OU Health/ Sarah Cannon Research Institute, Oklahoma City, Oklahoma
- Canada (3):
  - BC Cancer Center, Vancouver, British Columbia
  - University health Network (UHN)-University of Toronto, Toronto, Ontario
  - McGill University Health Care, Montreal, Quebec
- Spain (7):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Clinic de Barcelona Servicio de Oncología, Esc. 2, Planta 5 dcha, Barcelona, Catalonia
  - Hospital Universitario Quirón-Dexeus Servicio de Oncologia Médica, Barcelona
  - Hospital Universitario Dr. Josep Trueta - ICO de Girona, Servicio de Oncología Av. Francia s/n, Girona
  - Hospital Universitari Vall D Hebron, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz START Madrid-FJD- Unidad de Ensayos Fase I, Madrid
  - Hospital Universitario Virgen de la Arrixaca. Servicio de Oncología Ctra. Madrid-Cartagena, s/n, Murcia
- United Kingdom (6):
  - Lancashire Teaching Hospitals NHS Foundation Trust, Preston, Lancashire
  - Guy's & St Thomas' NHS Foundation Trust, London
  - The Royal Marsden NHS Foundation Trust, London
  - University College London Hospitals NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - The Royal Marsden NHS Foundation Trust, Sutton

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Dose escalation was limited to a single dose level for SL-172154 within each arm (in combination with the standard dose of PLD or MIRV). No participants were enrolled in other dose levels in either arm.
Groups:
- Pegylated Liposomal Doxorubicin + SL-172154: 3.0 mg/kg SL-172154 on Days 8 and 15 of every 28-day cycle plus pegylated liposomal doxorubicin (PLD) 40 mg/m2 on Day 1 of every 28-day cycle
- Mirvetuximab + SL-172154: 3.0 mg/kg SL-172154 on Days 8 and 15 of every 21-day cycle plus mirvetuximab (MIRV) 6.0 mg/kg on Day 1 of every 21-day cycle
Period: Overall Study
Arm/Group | Pegylated Liposomal Doxorubicin + SL-172154 | Mirvetuximab + SL-172154
Started | 21 | 65
Completed | 21 | 65
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pegylated Liposomal Doxorubicin + SL-172154: 3.0 mg/kg SL-172154 on Days 8 and15 of every 28-day cycle plus pegylated liposomal doxorubicin (PLD) 40 mg/m2 on Day 1 of every 28-day cycle
- Total: Total of all reporting groups
Arm/Group | Pegylated Liposomal Doxorubicin + SL-172154 | Mirvetuximab + SL-172154 | Total
Number analyzed (Participants) | 21 | 65 | 86
Age, Continuous [Median (Full Range); unit: years] | 58 [40 to 83] | 64 [44 to 80] | 64 [40 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 65 | 86
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 18 | 58 | 76
  Unknown or Not Reported | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 20 | 58 | 78
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: Participants]
  United States | 7 | 6 | 13
  Canada | 3 | 22 | 25
  United Kingdom | 6 | 13 | 19
  Spain | 5 | 24 | 29

OUTCOME MEASURES:

1. Primary Outcome: Evaluate Safety and Tolerability of SL-172154 When Administered With PLD or Mirvetixumab
Description: Number of participants with treatment emergent adverse events from dose escalation and expansion cohorts
Time Frame: From Day 1 to 30 days after last dose of SL-172154, PLD or Mirvetixumab, an average of approximately 6 months
Population: Subjects who received at least one dose of SL-172154, PLD or Mirvetixumab
Measure: Count of Participants; unit: Participants
Groups:
- Mirvetixumab + SL-172154: 3.0 mg/kg SL-172154 on Days 8 and15 of every 21-day cycle plus mirvetuximab (MIRV) 6.0 mg/kg on Day 1 of every 21-day cycle
Arm/Group | Pegylated Liposomal Doxorubicin + SL-172154 | Mirvetixumab + SL-172154
Number analyzed (Participants) | 21 | 65
Participants | 20 | 65

2. Secondary Outcome: To Assess Preliminary Evidence of Anti-tumor Activity of SL-172154 When Administered With PLD or Mirvetixumab
Description: Overall response rate per investigator assessment according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v 1.1)
Time Frame: approximately 24 months
Population: Response Evaluable Population
Measure: Count of Participants; unit: Participants
Groups:
- Mirvetixumab High (PS2+ ≥75%) + SL-172154; Mirvetixumab Low+Medium ((PS2+ ≥25% to <75%) + SL-172154: 3.0 mg/kg SL-172154 on Days 8 and15 of every 21-day cycle plus mirvetuximab (MIRV) 6.0 mg/kg on Day 1 of every 21-day cycle
Arm/Group | Pegylated Liposomal Doxorubicin + SL-172154 | Mirvetixumab High (PS2+ ≥75%) + SL-172154 | Mirvetixumab Low+Medium ((PS2+ ≥25% to <75%) + SL-172154
Number analyzed (Participants) | 20 | 39 | 26
Participants
  Complete response | 0 | 1 | 0
  Partial response | 4 | 12 | 4
  Stable Disease | 10 | 21 | 13
  Progressive Disease | 6 | 5 | 9
  Not Evaluable | 0 | 0 | 0

3. Secondary Outcome: Immunogenicity to SL-172154
Description: Number and proportion of participants with positive anti-drug antibody titer of those who were ADA negative at baseline
Time Frame: approximately 24 months
Population: Immunogenicity population.
Measure: Count of Participants; unit: Participants
Arm/Group | Pegylated Liposomal Doxorubicin + SL-172154 | Mirvetuximab + SL-172154
Number analyzed (Participants) | 20 | 60
Participants | 0 | 38

4. Secondary Outcome: Immunogenicity to MIRV
Description: Number and proportion of participants with positive anti-drug antibody titer of those who were ADA negative at baseline
Time Frame: approximately 24 months
Population: Immunogenicity population
Measure: Count of Participants; unit: Participants
Groups:
- Mirvetuximab + SL-172154: 3.0 mg/kg SL-172154 on Days 8 and15 of every 21-day cycle plus mirvetuximab (MIRV) 6.0 mg/kg on Day 1 of every 21-day cycle
Arm/Group | Mirvetuximab + SL-172154
Number analyzed (Participants) | 60
Participants | 8

5. Secondary Outcome: Maximum Serum Concentration (Cmax) of SL-172154
Description: The Cmax is the maximum observed serum concentration of SL-172154 following single and multiple doses
Time Frame: C1D8, C1D15, C2D8
Population: PK Population - number analyzed may be less than the number of participants in a given cohort if samples were below the limit of quantitation or not available for analysis
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Pegylated Liposomal Doxorubicin + SL-172154 | Mirvetuximab + SL-172154
Number analyzed (Participants) | 18 | 42
ng/mL
  C1D8: number analyzed (Participants) | 17 | 38
  C1D8 | 6022.23 (253.65) | 13248.42 (96.70)
  C1D15: number analyzed (Participants) | 11 | 34
  C1D15 | 13893.69 (90.44) | 8075.79 (97.53)
  C2D8: number analyzed (Participants) | 13 | 32
  C2D8 | 7083.44 (110.77) | 10375.13 (117.92)

6. Secondary Outcome: Area Under the Serum Concentration-time Curve (AUC) of SL-172154
Description: The AUC is the area under the serum concentration time curve of SL-172154 following single and multiple doses
Time Frame: C1D8, C1D15 and C2D8
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Pegylated Liposomal Doxorubicin + SL-172154 | Mirvetuximab + SL-172154
Number analyzed (Participants) | 18 | 42
h*ng/mL
  C1D8: number analyzed (Participants) | 17 | 38
  C1D8 | 9798.72 (239.36) | 27736.48 (79.72)
  C1D15: number analyzed (Participants) | 11 | 34
  C1D15 | 20157.25 (87.41) | 15324.37 (82.77)
  C2D8: number analyzed (Participants) | 13 | 31
  C2D8 | 11619.44 (132.43) | 21906.25 (116.59)

7. Secondary Outcome: Time at Which Maximum Concentration of SL-172154 is Observed (Tmax)
Description: The Tmax is the time at which the maximum concentration of SL-172154 is observed following single and multiple doses
Time Frame: C1D8, C1D15 and C2D8
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Groups:
- Pegylated Liposomal Doxorubicin +SL-172154: 3.0 mg/kg SL-172154 on Days 8 and 15 of every 28-day cycle plus pegylated liposomal doxorubicin (PLD) 40 mg/m2 on Day 1 of every 28-day cycle
Arm/Group | Pegylated Liposomal Doxorubicin +SL-172154 | Mirvetuximab + SL-172154
Number analyzed (Participants) | 18 | 42
hours
  C1D8: number analyzed (Participants) | 17 | 38
  C1D8 | 2.07 [1.9 to 4.1] | 2.22 [1.9 to 5.9]
  C1D15: number analyzed (Participants) | 11 | 34
  C1D15 | 2.15 [1.8 to 4.1] | 2.03 [1.8 to 4.5]
  C2D8: number analyzed (Participants) | 13 | 32
  C2D8 | 2.05 [1.1 to 4.4] | 2.28 [1.3 to 5.9]

8. Secondary Outcome: Maximum Serum Concentration (Cmax) of MIRV
Description: The Cmax is the maximum observed serum concentration of MIRV following single and multiple doses
Time Frame: Day 1 of each cycle, pre-dose and end of infusion (EOI)
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Mirvetuximab + SL-172154
Number analyzed (Participants) | 65
ng/mL
  C1D1 EOI: number analyzed (Participants) | 49
  C1D1 EOI | 137446.1 (15.8)
  C2D1 Predose: number analyzed (Participants) | 44
  C2D1 Predose | 3752.7 (54.7)
  C2D1- EOI: number analyzed (Participants) | 45
  C2D1- EOI | 121883.2 (71.5)
  C3D1-PREDOSE: number analyzed (Participants) | 34
  C3D1-PREDOSE | 4210.7 (49.9)
  C3D1-EOI: number analyzed (Participants) | 33
  C3D1-EOI | 122156.1 (61.7)
  C4D1-PREDOSE: number analyzed (Participants) | 28
  C4D1-PREDOSE | 3792.1 (74.4)
  C4D1-EOI: number analyzed (Participants) | 25
  C4D1-EOI | 125434.5 (16.1)
  C5D1-PREDOSE: number analyzed (Participants) | 21
  C5D1-PREDOSE | 4296.6 (55.4)
  C5D1-EOI: number analyzed (Participants) | 20
  C5D1-EOI | 130739.7 (14.3)
  C6D1-PREDOSE: number analyzed (Participants) | 14
  C6D1-PREDOSE | 4454.2 (58.8)
  C6D1-EOI: number analyzed (Participants) | 14
  C6D1-EOI | 117049.6 (11.5)
  C7D1-PREDOSE: number analyzed (Participants) | 10
  C7D1-PREDOSE | 3896.1 (64.2)
  C7D1-EOI: number analyzed (Participants) | 10
  C7D1-EOI | 103871.8 (16.0)
  C8D1-PREDOSE: number analyzed (Participants) | 6
  C8D1-PREDOSE | 5020.3 (40.6)
  C8D1-EOI: number analyzed (Participants) | 6
  C8D1-EOI | 108193.1 (13.3)
  C9D1-PREDOSE: number analyzed (Participants) | 4
  C9D1-PREDOSE | 4989.8 (50.1)
  C9D1-EOI: number analyzed (Participants) | 4
  C9D1-EOI | 105523.9 (16.4)
  C10D1-PREDOSE: number analyzed (Participants) | 3
  C10D1-PREDOSE | 3372.2 (116.3)
  C10D1-EOI: number analyzed (Participants) | 3
  C10D1-EOI | 105655.2 (11.2)
  C11D1-PREDOSE: number analyzed (Participants) | 2
  C11D1-PREDOSE | 5094.8 (19.0)
  C11D1-EOI: number analyzed (Participants) | 2
  C11D1-EOI | 99787.8 (11.2)

9. Primary Outcome: Establish the Recommended Phase 2 Dose (RP2D) for SL-172154 When Administered With PLD or Mirvetixumab
Description: Based on review of all data, including safety, tolerability, PK, antitumor activity, and PD effects"
Time Frame: From Day 1 to 30 days after last dose of SL-172154, PLD or Mirvetixumab, an average of approximately 6 months
Population: DLT evaluable population (Dose Escalation only)
Measure: Number; unit: mg/kg
Groups:
- Pegylated Liposomal Doxorubicin (PLD) + SL-172154: 3.0 mg/kg SL-172154 on Days 8 and15 of every 28-day cycle plus pegylated liposomal doxorubicin (PLD) 40 mg/m2 on Day 1 of every 28-day cycle
Arm/Group | Pegylated Liposomal Doxorubicin (PLD) + SL-172154 | Mirvetuximab + SL-172154
Number analyzed (Participants) | 8 | 7
mg/kg | 3.0 | 3.0

10. Secondary Outcome: Maximum Serum Concentration (Cmax) of Total Antibody (MIRV)
Description: The Cmax is the maximum observed serum concentration of Total Antibody (MIRV) following single and multiple doses
Time Frame: Day 1 of each cycle, pre-dose and end of infusion (EOI)
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Mirvetuximab + SL-172154
Number analyzed (Participants) | 65
ng/mL
  C1D1-EOI: number analyzed (Participants) | 49
  C1D1-EOI | 135716.4 (16.0)
  C2D1-PREDOSE: number analyzed (Participants) | 43
  C2D1-PREDOSE | 11901.6 (65.7)
  C2D1-EOI: number analyzed (Participants) | 45
  C2D1-EOI | 135856.9 (49.0)
  C3D1-PREDOSE: number analyzed (Participants) | 33
  C3D1-PREDOSE | 15986.7 (70.5)
  C3D1-EOI: number analyzed (Participants) | 33
  C3D1-EOI | 137898.7 (37.9)
  C4D1-PREDOSE: number analyzed (Participants) | 28
  C4D1-PREDOSE | 18388.2 (61.7)
  C4D1-EOI: number analyzed (Participants) | 25
  C4D1-EOI | 136454.6 (18.7)
  C5D1-PREDOSE: number analyzed (Participants) | 21
  C5D1-PREDOSE | 20115.1 (57.5)
  C5D1-EOI: number analyzed (Participants) | 20
  C5D1-EOI | 138756.5 (22.2)
  C6D1-PREDOSE: number analyzed (Participants) | 14
  C6D1-PREDOSE | 20283.3 (63.6)
  C6D1-EOI: number analyzed (Participants) | 14
  C6D1-EOI | 123020.4 (28.7)
  C7D1-PREDOSE: number analyzed (Participants) | 10
  C7D1-PREDOSE | 19007.7 (51.4)
  C7D1-EOI: number analyzed (Participants) | 10
  C7D1-EOI | 115087.0 (29.0)
  C8D1-PREDOSE: number analyzed (Participants) | 6
  C8D1-PREDOSE | 24546.8 (52.2)
  C8D1-EOI: number analyzed (Participants) | 6
  C8D1-EOI | 121205.9 (16.1)
  C9D1-PREDOSE: number analyzed (Participants) | 4
  C9D1-PREDOSE | 23604.6 (69.5)
  C9D1-EOI: number analyzed (Participants) | 4
  C9D1-EOI | 118301.1 (12.6)
  C10D1-PREDOSE: number analyzed (Participants) | 3
  C10D1-PREDOSE | 17972.6 (144.5)
  C10D1-EOI: number analyzed (Participants) | 3
  C10D1-EOI | 110207.7 (21.1)
  C11D1-PREDOSE: number analyzed (Participants) | 2
  C11D1-PREDOSE | 29331.9 (9.7)
  C11D1-EOI: number analyzed (Participants) | 2
  C11D1-EOI | 101638.6 (57.1)

11. Secondary Outcome: Maximum Serum Concentration (Cmax) of DM4 Payload and S-Methyl DM4 Payload (MIRV)
Description: The Cmax is the maximum observed serum concentration of DM4 Payload and S-Methyl DM4 payload following single and multiple doses
Time Frame: Day 1 of each cycle, pre-dose and end of infusion (EOI)
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- DM4 Payload; S-Methyl Payload: 3.0 mg/kg SL-172154 on Days 8 and15 of every 21-day cycle plus mirvetuximab (MIRV) 6.0 mg/kg on Day 1 of every 21-day cycle
Arm/Group | DM4 Payload | S-Methyl Payload
Number analyzed (Participants) | 65 | 65
ng/mL
  C1D1-EOI: number analyzed (Participants) | 49 | 50
  C1D1-EOI | 4.539 (40.775) | 0.191 (52.463)
  C2D1-PREDOSE: number analyzed (Participants) | 41 | 44
  C2D1-PREDOSE | 0.102 (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantitation | 0.798 (108.344)
  C2D1-EOI: number analyzed (Participants) | 44 | 43
  C2D1-EOI | 4.353 (48.036) | 3.228 (86.763)
  C3D1-PREDOSE: number analyzed (Participants) | 30 | 34
  C3D1-PREDOSE | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantitation | 0.711 (98.646)
  C3D1-EOI: number analyzed (Participants) | 31 | 34
  C3D1-EOI | 4.242 (45.189) | 2.712 (82.341)
  C4D1-PREDOSE: number analyzed (Participants) | 26 | 28
  C4D1-PREDOSE | 0.105 (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantitation | 0.645 (81.145)
  C4D1-EOI: number analyzed (Participants) | 26 | 26
  C4D1-EOI | 4.190 (39.346) | 2.336 (61.288)
  C5D1-PREDOSE: number analyzed (Participants) | 17 | 21
  C5D1-PREDOSE | 0.143 (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantitation | 0.513 (57.029)
  C5D1-EOI: number analyzed (Participants) | 20 | 21
  C5D1-EOI | 3.495 (49.810) | 1.812 (73.839)
  C6D1-PREDOSE: number analyzed (Participants) | 12 | 14
  C6D1-PREDOSE | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantitation | 0.565 (34.199)
  C6D1-EOI: number analyzed (Participants) | 14 | 14
  C6D1-EOI | 3.370 (38.460) | 1.963 (53.070)
  C7D1-PREDOSE: number analyzed (Participants) | 9 | 10
  C7D1-PREDOSE | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantitation | 0.500 (67.093)
  C7D1-EOI: number analyzed (Participants) | 10 | 9
  C7D1-EOI | 3.486 (55.862) | 1.460 (117.897)
  C8D1-PREDOSE: number analyzed (Participants) | 5 | 6
  C8D1-PREDOSE | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantitation | 0.736 (53.285)
  C8D1-EOI: number analyzed (Participants) | 4 | 6
  C8D1-EOI | 2.591 (29.962) | 2.238 (64.838)
  C9D1-PREDOSE: number analyzed (Participants) | 4 | 4
  C9D1-PREDOSE | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantitation | 0.526 (24.536)
  C9D1-EOI: number analyzed (Participants) | 3 | 4
  C9D1-EOI | 1.847 (30.813) | 1.438 (50.514)
  C10D1-PREDOSE: number analyzed (Participants) | 3 | 3
  C10D1-PREDOSE | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantitation | 0.700 (17.815)
  C10D1-EOI: number analyzed (Participants) | 3 | 3
  C10D1-EOI | 2.583 (74.475) | 1.599 (56.348)
  C11D1-PREDOSE: number analyzed (Participants) | 2 | 2
  C11D1-PREDOSE | NA (NA) — Not estimable based on subjects' concentration profiles, including values below the limit of quantitation | 0.728 (77.130)
  C11D1-EOI: number analyzed (Participants) | 2 | 2
  C11D1-EOI | 2.245 (9.463) | 1.544 (23.568)

ADVERSE EVENTS:
Time Frame: Subjects were followed continuously for all AEs starting when a subject signed the informed consent form, through 30 days after the last dose of SL-172154, PLD or Mirvetixumab, an average of approximately 6 months
Description: Serious Treatment-Emergent Adverse Events by Preferred Term
Groups:
- Pegylated Liposomal Doxorubicin + SL-172154: 3.0 mg/kg SL-172154 on Days 8 an15 of every 28-day cycle plus pegylated liposomal doxorubicin (PLD) 40 mg/m2 on Day 1 of every 28-day cycle
Arm/Group | Pegylated Liposomal Doxorubicin + SL-172154 | Mirvetuximab + SL-172154
All-Cause Mortality (participants affected / at risk) | 12/21 | 30/65
Serious Adverse Events (participants affected / at risk) | 4/21 | 17/65
Other Adverse Events (participants affected / at risk) | 20/21 | 65/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pegylated Liposomal Doxorubicin + SL-172154 (N=21) | Mirvetuximab + SL-172154 (N=65)
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 5
Ileus (Gastrointestinal disorders) | 1 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
General physical health deterioration (General disorders) | 0 | 2
Intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Cytokine release syndrome (Immune system disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Spinal cord infection (Infections and infestations) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Embolism (Vascular disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pegylated Liposomal Doxorubicin + SL-172154 (N=21) | Mirvetuximab + SL-172154 (N=65)
Nausea (Gastrointestinal disorders) | 11 | 32
Constipation (Gastrointestinal disorders) | 9 | 18
Abdominal pain (Gastrointestinal disorders) | 6 | 17
Diarrhoea (Gastrointestinal disorders) | 4 | 30
Stomatitis (Gastrointestinal disorders) | 6 | 4
vomiting (Gastrointestinal disorders) | 4 | 16
Abdominal distension (Gastrointestinal disorders) | 3 | 6
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 3
Dysphagia (Gastrointestinal disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 5
Dry mouth (Gastrointestinal disorders) | 0 | 5
Abdominal pain lower (Gastrointestinal disorders) | 0 | 4
Vision Blurred (Eye disorders) | 0 | 38
Dry eye (Eye disorders) | 0 | 20
Keratopathy (Eye disorders) | 0 | 19
Keratitis (Eye disorders) | 0 | 15
Photophobia (Eye disorders) | 0 | 9
Eye Pain (Eye disorders) | 0 | 6
Visual acuity reduced (Eye disorders) | 0 | 6
Visual impairment (Eye disorders) | 0 | 6
Cataract (Eye disorders) | 0 | 5
Vitreous floaters (Eye disorders) | 2 | 4
Fatigue (General disorders) | 9 | 26
Mucosal inflammation (General disorders) | 2 | 0
Oedema peripheral (General disorders) | 2 | 2
Non-cardiac chest pain (General disorders) | 0 | 8
Pyrexia (General disorders) | 2 | 3
Asthenia (General disorders) | 1 | 16
Chills (General disorders) | 0 | 4
Neutropenia (Blood and lymphatic system disorders) | 9 | 9
Anaemia (Blood and lymphatic system disorders) | 6 | 15
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 20
Lymphopenia (Blood and lymphatic system disorders) | 2 | 2
Folliculitis (Infections and infestations) | 2 | 0
Tooth infection (Infections and infestations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 2
Vulvovaginal candidiasis (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 6
COVID-19 (Infections and infestations) | 0 | 5
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 6 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Decreased appetite (Metabolism and nutrition disorders) | 6 | 12
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 11
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 13
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 6
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 5
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 4
Headache (Nervous system disorders) | 4 | 15
Dizziness (Nervous system disorders) | 2 | 6
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 26
Dysgeusia (Nervous system disorders) | 0 | 4
Neurotoxicity (Nervous system disorders) | 0 | 4
Infusion related reaction (Injury, poisoning and procedural complications) | 5 | 38
Alanine aminotransferase increased (Investigations) | 2 | 31
Aspartate aminotransferase increased (Investigations) | 2 | 30
Blood alkaline phosphatase increased (Investigations) | 1 | 5
Blood lactate dehydrogenase increased (Investigations) | 0 | 4
Weight decreased (Investigations) | 1 | 4
Embolism (Vascular disorders) | 2 | 0
Tachycardia (Cardiac disorders) | 0 | 4
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 4
Insomnia (Psychiatric disorders) | 0 | 6
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site agrees not to publish any Study Results or data before the publication of results from the Overall Study. After Sponsor has published the results of the Overall Study, Site may publish or present results generated at Site. If Sponsor has not published results of the Overall Study within 18 months of data base lock, Site may publish the results of the Study that were generated at Site. Site agrees to first submit to Sponsor the proposed publication at least 30 days prior to the submission.

DOCUMENTS (2):
  • Study Protocol (2024-06-25): https://cdn.clinicaltrials.gov/large-docs/33/NCT05483933/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-05): https://cdn.clinicaltrials.gov/large-docs/33/NCT05483933/SAP_001.pdf